CLINICAL TRIAL: NCT04796467
Title: A Pilot Prospective Comparison of 68Ga-P16-093 and 68Ga-PSMA-617 in the Same Group of Prostate Cancer Patients
Brief Title: 68Ga-P16-093 and 68Ga-PSMA-617 PET/CT Imaging in the Same Group of Prostate Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHPSMA093
Record Dates: First submitted 2021-02-23; First posted 2021-03-12 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA617 and 68Ga-P16-093 PET/CT scan (Experimental): Patients of Prostate cancer PET/CT imaging: In two consecutive days each patient underwent a PET/CT scan after intravenous administration of 68Ga-PSMA617 and 68Ga-P16-093, respectively.
  Interventions: Drug: 68Ga-PSMA-617; Drug: 68Ga-P16-093

INTERVENTIONS:
Drug: 68Ga-PSMA-617 — Intravenous injection of one dosage of 148-185 MBq (4-5 mCi) 68Ga-PSMA-617. Tracer doses of 68Ga-PSMA-617 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: 68Ga-PSMA-617 injection
Drug: 68Ga-P16-093 — Intravenous injection of one dosage of 148-185 MBq (4-5 mCi) 68Ga-P16-093. Tracer doses of 68Ga-P16-093 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: 68Ga-P16-093 injection

SUMMARY:
Prostate-specific membrane antigen (PSMA)-targeted PET imaging with 68Ga-labeled compounds is able to provide superior sensitivity and specificity to detect primary prostate tumor and its metastases, like the widely studied 68Ga-PSMA-617. This pilot study was prospectively designed to evaluate the early dynamic distribution of 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, which was compared with 68Ga-PSMA-617 in the same group of prostate cancer patients.

DETAILED DESCRIPTION:
Prostate cancer (PC) is one of the most common malignancies worldwide in men, with persistently high numbers dying from this disease. Due to low levels of glycolysis in prostate cancer cell, the uses of 18F-FDG PET/CT to detect prostate cancer and its metastases are limited. Prostate specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. Various low molecular weight radiopharmaceuticals targeting PSMA such as PSMA-617, PSMA-11 for 68Ga-labeling have been developed. 68Ga-PSMA PET/CT has demonstrated desirable sensitivity and specificity in the detection of prostate cancer lesions, which can find many micro lesions that cannot be identified by CT, MRI and bone scan. 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, with the urea fragment of a conjugate that employs the HBED-CC chelator for labeling with 68Ga(III). The HBED-based chelating ligand binds the 68Ga3+ ion with high affinity in a pseudo-octahedral N2O4 coordination sphere by its two phenolate O, two amino-acetate carboxylate O, and two amino N donor atoms. Mark A. Green et.al had demonstrated that 68Ga-P16-093 provided diagnostic information that appeared equivalent to 68Ga-PSMA-11 in prostate cancer patients presenting with biochemical recurrence, and 68Ga-P16-093 exhibits less urinary excretion than observed for 68Ga-PSMA-11. This pilot study was prospectively designed to evaluate the early dynamic distribution of 68Ga-P16-093 compared with 68Ga-PSMA-617 in the same group of prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated prostate cancer patients;
* 68Ga-PSMA617 and 68Ga-P16-093 PET/CT within two consecutive days;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic parameters | through study completion, an average of 1 year]
  the early dynamic distribution (SUVmax in tumor lesions and SUVmean in normal organs at different time points) of 68Ga-P16-093 in comparison with 68Ga-PSMA-617 in the same group of prostate cancer patients.

SECONDARY OUTCOMES:
detection capability of tumor | through study completion, an average of 1 year
  the tumor number detected by 68Ga-P16-093 PET/CT for prostate cancer in comparison with 68Ga-PSMA-617 PET/CT
SUVmax of tumor | through study completion, an average of 1 year
  the tumor uptake on 68Ga-P16-093 PET/CT for prostate cancer in comparison with 68Ga-PSMA-617 PET/CT

OTHER OUTCOMES:
PSMA expression and SUV | through study completion, an average of 1 year
  Correlation between PSMA expression and SUV in PET

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang G, Li L, Zang J, Hong H, Zhu L, Kung HF, Zhu Z. Head-to-Head Comparison of 68 Ga-P16-093 and 68 Ga-PSMA-617 PET/CT in Patients With Primary Prostate Cancer : A Pilot Study. Clin Nucl Med. 2023 Apr 1;48(4):289-295. doi: 10.1097/RLU.0000000000004566. Epub 2023 Jan 20. PMID 36727866
- [Derived] Wang G, Hong H, Zang J, Liu Q, Jiang Y, Fan X, Zhu Z, Zhu L, Kung HF. Head-to-head comparison of [68 Ga]Ga-P16-093 and [68 Ga]Ga-PSMA-617 in dynamic PET/CT evaluation of the same group of recurrent prostate cancer patients. Eur J Nucl Med Mol Imaging. 2022 Feb;49(3):1052-1062. doi: 10.1007/s00259-021-05539-1. Epub 2021 Sep 23. PMID 34557930